CLINICAL TRIAL: NCT06753877
Title: Clinical Monitoring of Individuals With Stroke During Inpatient Rehabilitation Using ICF:A Short-Term Follow-Up Study
Brief Title: Clinical Monitoring Using ICF
Acronym: ICF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Leyla Kaya Ozturk, Principal Investigator, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HÜ-OT-LKO-02
Record Dates: First submitted 2024-12-23; First posted 2024-12-31 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Stroke
Keywords: stroke; activities of daily living; participation; rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: One group was investigated within the ICF framework
Masking Description: The therapist who conducted the assessment tests was unaware of the study design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aspirin (single group) (Experimental): The present study has one group. Holistic rehabilitation service was provided to all individuals. The program involved different therapies. Participants were given standard physiotherapy services (electrotherapy, exercise, gait training, hydrotherapy, respiratory therapy) and standard occupational therapy services. Occupational therapy interventions were provided by the researchers.
  Interventions: Behavioral: holistic rehabilitation

INTERVENTIONS:
Behavioral: holistic rehabilitation — Holistic rehabilitation service All participants in the study were cared for in the inpatient unit. The same physician and nurses followed the participants for 1 month. The participants were regularly taking their medication and had no co-morbidities. All participants stayed in double rooms and all stayed with their caregivers. The assessments were carried out within the first 3 days of admission to the inpatient unit. The second assessments were repeated by the same professional. Rehabilitation interventions were provided by different therapists. Participants were given standard physiotherapy services (electrotherapy, exercise, gait training, hydrotherapy, respiratory therapy) and standard occupational therapy services. Occupational therapy interventions were provided by the researchers. Physiotherapy services were provided by physiotherapists working full-time in the hospital. Physiotherapy was provided 5 days a week and occupational therapy was provided 3 days a week.

SUMMARY:
The present study examined stroke patients who applied to occupational therapy units within the framework of ICF, following the rehabilitation process, and defining frequently used measurements in terms of ICF codes

DETAILED DESCRIPTION:
The International Classification of Functioning (ICF) is a standardized method frequently used by health professionals. This follow-up study was performed in accordance with the Declaration of Helsinki. The present study examined stroke patients who applied to occupational therapy units within the framework of ICF, following the rehabilitation process, and defining frequently used measurements in terms of ICF codes. Participants were recruited from the patients who applied to the Occupational Therapy Clinic of Etlik City Hospital. Participants who agreed to participate in the study signed an informed consent form. First, the scales were defined within the framework of ICF. Individuals who had a stroke and were hospitalized in the Physiotherapy and Rehabilitation Clinic of Etlik City Hospital and included in the study were evaluated using ICF parameters within the first 3 days of their hospitalization. All individuals were given a holistic rehabilitation program. Individuals who received inpatient treatment and stayed in the hospital for one month were re-evaluated. Other individuals who were not included in the study benefited from traditional inpatient treatment services. Upon evaluating the rehabilitation service within the framework of ICF, significant changes were observed in body functions, activity, and participation. It is recommended that ICF be used by occupational therapists and other health professionals, that the scales be associated with ICF codes, and that holistic rehabilitation services be developed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stroke, age between 18 and 64 years,
* Being served by hospital, being enrolled in the occupational therapy,
* Volunteering to participate in the study

Exclusion Criteria:

* Individuals with orthopedic, psychological or neurological conditions other than stroke that could affect their functioning and those with moderate or severe aphasia were not included in the study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Functional Independence Scale (FIM) | 1 month
  The FIM is a scale that measures a person's level of independence in basic motor and cognitive activities of daily living. It consists of 18 items and assesses 2 sub-areas. 1) motor function and 2) cognitive function. Each item is scored on a detailed scale ranging from 1 to 7 (level 1 = fully dependent, level 7 = fully independent). The total score ranges from 18 to 126. The higher the person's score, the higher the level of independence (Ravaud et al., 1999). The Turkish cultural adaptation study was conducted.

SECONDARY OUTCOMES:
Mini Mental State Examination (MMSE) | 1 month
  The MMSE, which assesses cognitive impairment, is a scale developed. It is a useful, short and standardised tool that can be used to determine cognitive level. It consists of five main sections: orientation, registration, attention and calculation, recall, and language with a total of eleven items. The score range is 0-30. A higher score indicates a higher cognitive level. The Turkish validity and reliability were carried out.

OTHER OUTCOMES:
Stroke Impact Scale version 3.0 (SIS v-3.0): | 1 month
  The SIS is a scale designed to assess clients' perceived quality of life after stroke. The scale was developed as SIS 2.0 and updated to SIS 3.0. It consists of 8 domains (strength, hand function, mobility, ADL/IADL, memory and thinking, communication, emotion, and social participation) and 59 questions. The degree of difficulty with activities in the past week is rated on a 5-point Likert scale. The score for each domain ranges from 0 to 100. In addition to the 8 sub-sections, the perception of recovery after stroke is assessed using a 0-100 point visual analog scale (0: no recovery, 100: full recovery). The Turkish validity and reliability study was conducted.
Lawton-Brody Instrumental Activities of Daily Living (Lawton-Brody IADL) | 1 month
  This test, which measures the subjective level of independence in IADL, was developed. It consists of 8 questions about "ability to use phone, shopping, food preparation, housekeeping, laundry, mode of transportation, responsibility for own medications, ability to handle finances". It is scored on a 0-8 scale, with a low score indicating high dependency. The Turkish cultural adaptation study was conducted.
Frenchay Activities Index (FAI): | 1 month
  The Frenchay Activities Index (FAI) is a scale designed to assess the activities of daily living and social participation of individuals. It consists of 15 items asking how often activities of daily living, such as preparing meals and washing up, and activities of social participation, such as socialising and driving, are performed. The first 10 items express the frequency of activities performed in the last three months and the remaining items express the frequency of activities performed in the last six months. Each item consists of a 4-point Likert scale (0=never, 3=at least once a week) and the total score ranges from 0 (not active) to 45 (very active). The Turkish cultural adaptation study was conducted.

CONTACTS AND LOCATIONS:
Overall Officials: leyla kaya öztürk, MSc, Principal Investigator — Mardin Training and Research Hospital
Locations (1):
- Mardin Traning and Rsearch Hospital, Mardin, Artuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No